CLINICAL TRIAL: NCT06010862
Title: A Safety and Efficacy Clinical Study of CEA-targeted CAR-T Therapy forCEA-positive Advanced/Metastatic Malignant Solid Tumors
Brief Title: Clinical Study of CEA-targeted CAR-T Therapy for CEA-positive Advanced/Metastatic Malignant Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Collaborators: The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBC051
Record Dates: First submitted 2023-08-18; First posted 2023-08-25 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-08

CONDITIONS: Gastric Cancer; Colon Cancer; Pancreas Cancer; Esophagus Cancer; Cholangiocarcinoma; Lung Cancer; Breast Cancer
Keywords: CAR-T; CEA
MeSH Terms: conditions — Stomach Neoplasms; Colonic Neoplasms; Pancreatic Neoplasms; Esophageal Neoplasms; Cholangiocarcinoma; Lung Neoplasms; Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous of CEA-targeted CAR-T (Experimental): Infusion of CEA-targeted CAR-T cells by dose of 1-10x106 cells/kg
  Interventions: Biological: CEA CAR-T cells
- intraperitoneal injection of CEA-targeted CAR-T (Experimental): Infusion of CEA-targeted CAR-T cells by dose of 1-10x106 cells/kg
  Interventions: Biological: CEA CAR-T cells

INTERVENTIONS:
Biological: CEA CAR-T cells — After lymphodepletion with Fludarabine and Cyclophosphamide,CAR T cells were transfused intravenically
  Arms: Intravenous of CEA-targeted CAR-T
Biological: CEA CAR-T cells — After lymphodepletion with Fludarabine and Cyclophosphamide,CAR T cells were injected intraperitoneally
  Arms: intraperitoneal injection of CEA-targeted CAR-T

SUMMARY:
This is a phase I clinical study to evaluate the safety and tolerability of CAR-T in patients with CEA-positive advanced/metastatic solid tumors, and to obtain the maximum tolerated dose of CAR-T and phase II Recommended dose.

DETAILED DESCRIPTION:
This is a single-center, double-arm, open-label study. The study plans to set up 2 groups,Intravenous infusion group have 4 dose groups, adopting a dose-escalating 3+3 design, and plan to recruit about 12 subjects with CEA-positive advanced/metastatic solid tumors.Intraperitoneal injection group have 4 dose groups, adopting a dose-escalating 3+3 design, and plan to recruit about 12 subjects with CD70-positive advanced/metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, male or female;
2. Advanced, metastatic or recurrent malignant tumors diagnosed by histology or pathology, mainly colorectal cancer, esophageal cancer, gastric cancer, and pancreatic cancer;
3. After receiving at least second-line standard treatment failure (disease progression or intolerance, such as surgery, chemotherapy, radiotherapy, etc.) or lack of effective treatment methods;
4. Immunohistochemical staining of tumor samples within 3 months confirmed that the tumor was CEA positive (clear membrane staining, positive rate ≥ 10%); , the positive rate ≥ 10%), the serum CEA of the patient is required to exceed 10ug/L.
5. At least one assessable lesion according to RECIST 1.1 criteria;
6. ECOG score 0-2 points;
7. No serious mental disorder;
8. Unless otherwise specified, the function of the vital organs of the subject shall meet the following conditions:

   1. Blood routine: white blood cells>3.0×10^9/L, neutrophils>0.8×10^9/L, lymphocytes cells>0.5×10^9/L, platelets>75×10^9/L, hemoglobin>80g/L;
   2. Cardiac function: echocardiography showed cardiac ejection fraction ≥50%, and no obvious abnormality was found on electrocardiogram;
   3. Renal function: serum creatinine≤2.0×ULN;
   4. Liver function: ALT and AST ≤3.0×ULN (for patients with liver tumor infiltration, it can be relaxed to ≤5.0×ULN);
   5. Total bilirubin≤3.0×ULN;
   6. Oxygen saturation ≥95% in non-oxygen state.
9. Have apheresis or venous blood collection standards, and have no other contraindications for cell collection;
10. Subjects agree to use reliable and effective contraceptive methods for contraception within 1 year after signing the informed consent form to receiving CAR-T cell infusion (excluding rhythm contraception);
11. The patients themselves or their guardians agree to participate in this clinical trial and sign the ICF, indicating that they understand the purpose and procedures of this clinical trial and are willing to participate in the research.

Exclusion Criteria:

1. Those who have central nervous system metastasis or meningeal metastasis at the time of screening are judged by the investigator to be unsuitable for inclusion;
2. Participated in other clinical studies within 1 month before screening;
3. vaccinated with live attenuated vaccine within 4 weeks before screening;
4. Received the following anti-tumor treatments before screening: Received chemotherapy, targeted therapy or other experimental drug treatments within 14 days or at least 5 half-lives (whichever is shorter);
5. Active infection or uncontrollable infection requiring systemic treatment;
6. Patients with intestinal obstruction, active gastrointestinal bleeding, or a history of gastrointestinal bleeding within 3 months;
7. Except for alopecia or peripheral neuropathy, the toxicity of previous anti-tumor therapy has not improved to the baseline level or ≤ grade 1;
8. Suffering from any of the following heart diseases:

   1. New York Heart Association (NYHA) stage III or IV congestive heart failure;
   2. Myocardial infarction or coronary artery bypass grafting (CABG) within 6 months before enrollment;
   3. Clinically significant ventricular arrhythmia, or a history of unexplained syncope (except those caused by vasovagal or dehydration);
   4. History of severe non-ischemic cardiomyopathy;
9. Patients with active autoimmune disease, or other patients requiring long-term immunosuppressive therapy;
10. Suffering from other uncured malignant tumors in the past 3 years or at the same time, except cervical carcinoma in situ and basal cell carcinoma of the skin;
11. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA titer test is greater than the normal range; hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C Virus (HCV) RNA test is greater than the normal range; human immunodeficiency virus (HIV) antibody positive; syphilis test positive;
12. Women who are pregnant or breastfeeding;
13. Other investigators deem it unsuitable to participate in the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-09-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse events after CEA CAR-T cells infusion [Safety and Tolerability] | 28 days
  Therapy-related adverse events were recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0)
Obtain the maximum tolerated dose of CEA CAR-T cells[Safety and Tolerability] | 28 days
  Dose-limiting toxicity after cell infusion

SECONDARY OUTCOMES:
Disease control rate of CAR-T cell preparations in CEA positive advanced malignancies [Effectiveness] | 3 months
  Disease control rate: The proportion of subjects who achieved CR, PR, SD after treatment accounted for all treated subjects (Assessed based on RECIST criteria)，the minimum value is 0%，maximum value is 100%, and higher scores mean a better outcome.
Objective response rate (ORR) of CEA CAR-T treatment in patients with CD70-positive advanced malignancies[Effectiveness] | 3 months
  Objective response rate includes：The proportion of subjects who achieved CR, PR after treatment accounted for all treated subjects (Assessed based on RECIST criteria)，the minimum value is 0%，maximum value is 100%, and higher scores mean a better outcome.
Duration of Response (DOR) of CEA CAR-T treatment in patients with CEA-positive advanced malignancies[Effectiveness] | 3 months
  DOR will be assessed from the first assessment of CR/PR/SD to the first assessment of recurrence or progression of the disease or death from any cause
Overall survival(OS)of CEA CAR-T treatment in patients with CEA-positive advanced malignancies[Effectiveness] | 2 years
  OS will be assessed from the first CEA-CAR-T cell infusion to death from any cause (Assessed based on RECIST criteria)
Progress-free survival(PFS) of CEA CAR-T treatment in patients with CD70-positive advanced malignancies[Effectiveness] | 2 years
  PFS will be assessed from the first CEA-CAR-T cell infusion to death from any cause or the first assessment of progression(Assessed based on RECIST criteria)
AUCS of CEA CAR-T cells [Cell dynamics] | 3 months
  AUCS is defined as the area under the curve in 90 days
CMAX of CEA CAR-T cells [Cell dynamics] | 3 months
  CMAX is defined as the highest concentration of CEA CAR-T cells expanded in
TMAX of CEA CAR-T cells[Cell dynamics] | 3 months
  TMAX is defined as the time to reach the highest concentration
Pharmacodynamics of CEA CAR-T cells[Cell dynamics] | 3 months
  Concentration levels of CAR-T-related serum cytokines such as CRP, IL-6, ferritin at each time point

OTHER OUTCOMES:
The correlation between CEA positive rate and safety | 2 years
  assessment the correlation between CEA positive rate and the incidence of CRA and ICANS
Correlation between CEA positive rate and efficacy | 2 years
  assessment the correlation between CEA positive rate and the disease control rate，Disease control rate: including CR, PR and SD
Overall survival(OS)of CEA CAR-T treatment in patients with CEA-positive advanced malignancies[Effectiveness] | 2 years
  OS will be assessed from the first CEA-CAR-T cell infusion to death from any cause (Assessed by investigators based on IRECIST criteria)
Progress-free survival(PFS) of CEA CAR-T treatment in patients with CEA-positive advanced malignancies[Effectiveness] | 2 years
  PFS will be assessed from the first CEA-CAR-T cell infusion to death from any cause or the first assessment of progression (Assessed by investigators based on IRECIST criteria)
Duration of Response (DOR) of CEA CAR-T treatment in patients with CEA-positive advanced malignancies[Effectiveness] | 2 years
  DOR will be assessed from the first assessment of CR/PR/SD to the first assessment of recurrence or progression of the disease or death from any cause (Assessed by investigators based on IRECIST criteria)

CONTACTS AND LOCATIONS:
Overall Officials: Fei Li, M.D, Principal Investigator — The First Affiliated Hospital of Nanchang University
Locations (1):
- The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China